CLINICAL TRIAL: NCT00577044
Title: Non Alcoholic Fatty Liver Disease (NAFLD) in Hong Kong: Natural History and Development of Liver Complications
Brief Title: Non Alcoholic Fatty Liver Disease (NAFLD) in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Other Study IDs: UW 05-120 T/783; HARECCTR0500006; KW/EX/05-036
Record Dates: First submitted 2007-07-06; First posted 2007-12-19 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-06

CONDITIONS: Fatty Liver
Keywords: NAFLD
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

SUMMARY:
The true incidence and prevalence of NAFLD in Hong Kong has not been determined. The natural history of NAFLD is not well defined partly because of differences in the exclusion limit of alcohol and the required histological criteria between studies. NAFLD is previously believed to be a benign non-progressive condition, but it has since been determined that a subset of patients can progress to cirrhosis and even hepatocellular carcinoma.

In fact in a recent histological review of NAFLD, fibrosis or liver cirrhosis was present in 15-50% of patients at index liver biopsy. The presence of obesity or type 2 diabetes mellitus are the strongest predictors of fibrosis. These same risk factors are also more common in patients with cryptogenic cirrhosis. Further evidence of the link between diabetes, obesity and NAFLD are mainly from the field of liver transplantation. In patients who underwent liver transplantation for cryptogenic liver cirrhosis, NAFLD recuured in a quarter of the hepatic allografts. The patients with recurrent NAFLD were more likely to be diabetic and had a higher body mass index (BMI) at the time of recurrent NAFLD. This suggests that NAFLD may have a significant role in the pathogenesis of crytogenic cirrhosis.

Although NAFLD was initially described as a slowly progressive disease, there are emerging data which shows that it can progress rapidly. Liver failure has even been described in patients with NAFLD after bariatric surgery, and a recent report described 5 cases of subacute liver failure in obese middle aged females with NAFLD related cirrhosis. NAFLD can also affect the progression of other diseases as well. Hepatic steatosis related to visceral obesity is a major independent risk factor for fibrogenesis related to chronic HCV hepatitis.

However, the prevalence of NAFLD and its interaction with chronic HBV, if any, is uncertain. This study aims to determine the prevalence of NAFLD in patients with unknown cause of hepatitis and to determine the histological fibrosis and inflammation in chronic HBV patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Gender: male and female

Exclusion Criteria:

* HBV patients and fatty liver HCV HIV

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2004-06; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: George K Lau, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (5):
- China (5):
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Department of Pathology, Princess Margaret Hospital, Hong Kong
  - Department of Pathology, Queen Elizabeth Hospital, Hong Kong
  - Department of Pathology, Queen Mary Hospital, Hong Kong
  - Department of Pathology, Tuen Mun Hospital, Hong Kong